CLINICAL TRIAL: NCT01302171
Title: Randomised Controlled Trial to Compare the Effects of G-CSF (Granocyte™) and Autologous Bone Marrow Progenitor Cells on Quality of Life and Left Ventricular Function in Patients With Idiopathic Dilated Cardiomyopathy
Brief Title: Bone Marrow Derived Adult Stem Cells for Dilated Cardiomyopathy
Acronym: REGEN-DCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); University College London Hospitals (Other)
Responsible Party: Principal Investigator, Anthony Mathur, Clinical and Research Lead (Cardiology), Barts & The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-013112-12
Record Dates: First submitted 2011-02-21; First posted 2011-02-24 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Dilated Cardiomyopathy
Keywords: dilated cardiomyopathy; adult stem cells; bone marrow progenitor cells; bone marrow stem cells; autologous; granulocyte-colony stimulating factor; intracoronary injection; left ventricular function; To determine if patient's own bone marrow derived stem cells can be used to improve cardiac function
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Granulocyte Colony-Stimulating Factor; Lenograstim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peripheral (Experimental): Half the patients will be randomised to the non-interventional part of the trial. In this subgroup of patients will be randomised 1:1 to 5 day course of subcutaneous placebo injections or a 5 day course of G-CSF(Granocyte™) subcutaneous injections
  Interventions: Drug: granulocyte colony stimulating factor (GCSF)
- Interventional arm (Experimental): In the subgroup of the interventional arm patients will be randomised 1:1 to receive a 5 day course of subcutaneous G-CSF (Granocyte™) injections and bone marrow aspiration at day 5, they will then receive either stem cells or placebo via intracoronary injection
  Interventions: Procedure: bone marrow mononuclear cells

INTERVENTIONS:
Drug: granulocyte colony stimulating factor (GCSF) — 10mcg/kg per day 5 days
  Other Names: Lenograstim, Granocyte™, Chugai Pharma UK, Limited
  Arms: Peripheral
Procedure: bone marrow mononuclear cells — intra coronary injection of stem cells or placebo
  Arms: Interventional arm

SUMMARY:
A randomised, double-blind, placebo-controlled trial to evaluate the role of intracoronary injection of progenitor cells compared to placebo injection in patients with Dilated Cardiomyopathy who have been pre-treated with G-CSF (Granocyte™) injections for 5 days, and patients treated with a 5 day course of G-CSF (Granocyte™) injection only compared to placebo injection

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with a confirmed diagnosis of dilated cardiomyopathy (NYHA II-III) attending their local 'Heart Failure clinic' who are on optimal heart failure treatment, under supervision from their physician or heart failure nurse specialist, and have no other treatment options
* Patients who are NYHA II that have been hospitalised with a dilated cardiomyopathy related condition
* Coronary angiography will be performed where necessary to confirm the diagnosis and ensure no other conventional treatment options are indicated
* Prior to recruitment to the study patients at risk of ventricular arrhythmia will have undergone electrophysiological assessment and appropriate clinical management (including implantable defibrillator insertion) where indicated (as per NICE guidelines)

Exclusion Criteria:

* NYHA I
* Referral hospitals most recent documented ejection fraction of >45% (any imaging modality)
* The presence of cardiogenic shock
* The presence of acute left and/or right sided pump failure as judged by the presence of pulmonary oedema and/or new peripheral oedema
* Known severe pre-existent left ventricular dysfunction (with a documented ejection fraction of <10% from referral hospital) prior to randomisation
* Congenital cardiac disease
* Cardiomyopathy secondary to a reversible cause that has not been treated e.g. thyroid disease, alcohol abuse, hypophosphataemia, hypocalcaemia, cocaine abuse, selenium toxicity & chronic uncontrolled tachycardia
* Cardiomyopathy in association with a neuromuscular disorder e.g. Duchenne's progressive muscular dystrophy
* Previous cardiac surgery
* Contra-indication for bone marrow aspiration
* Known active infection
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), HTLV or syphilis.
* Chronic inflammatory disease requiring ongoing medication
* Serious known concomitant disease with a life expectancy of less than one year
* Follow-up impossible (no fixed abode, etc)
* Patients with an irregular heart rhythm (AF allowed if paced in a regular rhythm)
* Patients with renal impairment (Creatinine >200mmol/L)
* Neoplastic disease without documented remission within the past 5 years
* Weight>140kg
* Subjects of childbearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction as measured by cardiac magnetic resonance imaging or computerised tomography | 3 months

SECONDARY OUTCOMES:
Change in: Concentrations of N-terminal prohormone of brain natriuretic peptide (cardiac enzyme) | 3 months and 12 months
Changes in V02 max (exercise capacity) | 3 months and 12 months
Changes in left ventricular ejection fraction, ventricular dimensions as measured by cardiac magnetic resonance imaging or computerised tomography | 3 months and 12 months
Functional class changes according to NYHA and quality of life (QoL - EQ-5D & Kansas City) questionnaires | 3 months and 12 months
Occurrence of a Major Adverse Cardiac Event (MACE) defined as cardiac death, myocardial infarction (CK / CK-MB over 2 times the upper limit of normal) | 3 months and 12 months
Hospitalization for Heart failure & the occurrence of major arrhythmias defined as symptomatic ventricular tachycardia or survived sudden death | 3 months and 12 months
The occurrence of major arrhythmias defined by symptomatic ventricular tachycardia or survived sudden death | 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, MD FRCP FESC, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- London Chest Hospital, London, United Kingdom

REFERENCES:
- [Background] Arnous S, Mozid A, Mathur A. The Bone Marrow Derived Adult Stem Cells for Dilated Cardiomyopathy (REGENERATE-DCM) trial: study design. Regen Med. 2011 Jul;6(4):525-33. doi: 10.2217/rme.11.29. PMID 21749209